CLINICAL TRIAL: NCT01650974
Title: High Flow Nasal OXygen Therapy in High Risk Patients of Hypoxia Undergoing Diagnostic BRONCHOscopy: A Prospective, Randomized, Controlled Study
Brief Title: High Flow Nasal OXygen Therapy in High Risk Patients of Hypoxia Undergoing Diagnostic BRONCHOscopy
Acronym: HFNOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Young-Jae Cho, Seoul National University Bundang Hospital, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: E-1205-154-002; H-1206-074-414 (Other: Seoul National University Hospital)
Record Dates: First submitted 2012-07-24; First posted 2012-07-26 (Estimated); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Hypoxia
Keywords: high flow nasal oxygen therapy; diagnostic bronchoscopy
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- conventional oxygen therapy (No Intervention): conventional nasal prong with FiO2 ~0.4
- HFNOT (Experimental): high flow nasal oxygen therapy with starting FiO2 0.4 and Flow 40 L/min
  Interventions: Device: HFNOT
- sham-HFNOT (Sham Comparator): same device with FiO2 ~0.4, NO high flow
  Interventions: Device: HFNOT

INTERVENTIONS:
Device: HFNOT — high flow nasal oxygen therapy
  Other Names: high flow nasal oxygen therapy(OPTIFLOW)
  Arms: HFNOT; sham-HFNOT

SUMMARY:
The purpose of this study is to determine the efficacy and safety of nasal high flow oxygen therapy during diagnostic bronchoscopy.

DETAILED DESCRIPTION:
Hypoxemia is frequently seen during diagnostic bronchoscopy. Nasal prong or other existing oxygen supply methods are often difficult to maintain adequate oxygenation during bronchoscopy. In particular, bronchoscopy to patients already showing hypoxemia can be dangerous even though applying conventional oxygen therapy. Thus, we want to elucidate the usefulness of nasal high flow oxygen therapy to hypoxemic patients undergoing diagnostic bronchoscopy.

ELIGIBILITY:
Inclusion Criteria: 1 or 2

1. PaO2 < 60 mmHg on ABGA or SpO2 < 90 % in room air AND SpO2 ≥ 95% or PaO2 ≥ 75mmHg in low flow oxygen therapy
2. Planning to diagnostic bronchoscopic procedure (e.g. bronchial washing, BAL, bronchoscopic biopsy, EBUS-TBNA etc.)

Exclusion Criteria:

1. patients who did not agree to provide information
2. patients requiring for emergent intubation
3. patients can not wear or be already applied high flow nasal oxygen therapy
4. patients with unstable vital sign(e.g. severe hypotension, uncontrolled arrhythmia, etc.)
5. patients with multiple organ failures
6. patients with plan to therapeutic bronchoscopic procedure(e.g. intervention)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2012-07; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Success rate of bronchoscopy | 1 day
  Success is defined as completion of planned diagnostic procedure with the oxygen saturation or partial pressure of oxygen in arterial blood was similar to the level of before the procedure.
  Failure is defined as incompletion of planned diagnostic procedure due to sustained hypoxemia or else.
  Furthermore failure is defined as hypoxemia(SaO2 <88%) was developed more than 2 times even though planned procedure was completed.
Total duration of hypoxia | 1 day
  total duration of hypoxia(oxygen saturation ≤88%) during procedure or after procedure.

SECONDARY OUTCOMES:
frequency of hypoxia | 1 day
  frequency of hypoxia(oxygen saturation ≤88%) during procedure or after procedure.
switch to oxygen therapy method | 1 day
  Increase oxygen apply or change of oxygen therapy method to high flow system.
change of respiratory symptoms | 1 day
  scoring of dyspnea symptoms, patients comfort.

CONTACTS AND LOCATIONS:
Overall Officials: Young-Jae Cho, MD, MPH, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea